CLINICAL TRIAL: NCT07269938
Title: Mapping B-cell Biology Across the Cardiovascular Territories of Giant Cell Arteritis: Towards a New Therapeutic Approach (RituxiMAP GCA)
Acronym: RituxiMAP GCA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC25173
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Giant cell arteritis; Vasculitis; Rituximab; PET scanning
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LV-GCA group: Patients with a diagnosis of active, large vessel GCA
  Interventions: Diagnostic Test: Zirconium Zr 89 labelled rituximab
- AA control group: Patients with a diagnosis of atherosclerotic aortic aneurysm
  Interventions: Diagnostic Test: Zirconium Zr 89 labelled rituximab
- BCMID control group: Patients with a diagnosis of a B-cell mediated inflammatory disorder
  Interventions: Diagnostic Test: Zirconium Zr 89 labelled rituximab

INTERVENTIONS:
Diagnostic Test: Zirconium Zr 89 labelled rituximab — All participants will receive a PET scan with zirconium Zr-89 labelled rituximab. Those in the LV-GCA group will receive a follow-up scan after a period of treatment.

SUMMARY:
B cells are a component of the immune system which appear be important in causing all forms of cardiovascular disease. Until now, it has not been possible to directly study these cells in living patients (essential to assess their potential as the target of new treatments). For the first time in any cardiovascular disease, this study will apply cutting edge scanning technology to visualise B cells in the blood vessels of giant cell arteritis (GCA) patients. GCA is a common and potentially deadly disorder of the blood vessels which is caused by abnormalities of the immune system. Current treatments are mainly limited to steroids. Unfortunately, these drugs bring tremendous side effects and so there is an urgent requirement to discover alternatives.

Laboratory investigations tell us that B cells are highly present in GCA and so if the proposed scanning technology fails to identify these cells in the blood vessels of participants, then the technology is unlikely to be useful for other cardiovascular diseases. If, however, the study does successfully visualise B cells, this knowledge could pave the way for clinical trials of B cell targeted treatments (already established in other conditions) as steroid alternatives in GCA.

This study aims to map the distribution of the radiotracer zirconium-89 labelled rituximab within the blood vessels of patients with newly diagnosed GCA and compare this with two separate control groups without the condition. This will allow us to determine the role of B cells within this condition, and whether patients would benefit from B cell-depleting treatments such as rituximab.

DETAILED DESCRIPTION:
Giant cell arteritis (GCA) is an auto-immune condition which causes inflammation of medium and large arteries around the body. Previously thought to primarily affect the temporal arteries, there is now an understanding that the disease is more widespread, with most patients demonstrating involvement of the aorta and other large vessels.

Current treatments rely heavily on steroids which can cause significant side effects. Other novel treatments for GCA are also limited, with many patients relapsing once treatment is withdrawn. There is therefore an urgent need for new therapies for GCA, particular in those patients with large vessel involvement (LV-GCA)

B cells - a type of immune cell - are thought to play a key role in causing damage to blood vessels in diseases like atherosclerosis and may be implicated in GCA. Accordingly, a potential treatment approach may be to target B cells using a drug called rituximab (RTX), which is already used in other immune conditions. To explore this possibility safely and effectively, we need a way to see where B cells are in the body, and how they are affected by treatment in GCA. This can be achieved using total body PET scanning with zirconium-89-labeled rituximab.

By injecting patients with zirconium-89-labeled rituximab and then undergoing total body PET scanning, this study hopes to track B cells in real time within the blood vessels of those with GCA. This scan has been used safely in studies of cancer, lung disease, and rheumatoid arthritis.

In summary, the aim of this feasibility study is to:

* Map the location of B cells in those with LV-GCA
* Compare this activity with blood and biopsy samples
* Test whether steroid treatment reduces B cell activity

If successful, this could pave the way for B-cell targeting treatments (like rituximab) that reduce the need for steroids and better control inflammation in LV-GCA.

This will be an observational longitudinal pilot study with a nested baseline case-control comparison. The study will recruit 15 patients with LV-GCA from across Scotland. Participants will attend the University of Edinburgh for a baseline total body 89Zr-RTX PET/CT scan and then receive 4 months of steroid therapy. They will then complete the study with a final total body 89Zr-RTX PET/CT scan. The study will also recruit two control groups. The first will be a group of 10 participants with alternative B cell mediated immune disorders (BCMID group), including (but not limited to) systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis, myositis, and Sjogren's syndrome. The second group will include 5 participants with atherosclerosis associated aortic aneurysms. The BCMID control group will receive both baseline and follow-up scans. The AA control group will receive a baseline scan only. All participants will provide a blood sample at each visit in order to compare blood B cells with B cells pictured on the scan. If GCA patients have already had a biopsy of a blood vessel as part of their standard care, the investigators will compare tissue B cells with B cells pictured on the scan. If those in the AA group have any available aortic tissue which has previously been removed at time of aneurysm repair, the investigators will also seek to compare B cell populations within this tissue and on the scan.

As this is a pilot study, and 89Zr-RTX has not previously been used to image disease in GCA, the optimum time period between radiotracer injection and PET scan is not yet known. Accordingly, the first 5 participants in the GCA group will undergo PET scans and coupled blood tests at 3, 5 and 7 days after injection of the radiotracer. This will allow determination of the best time to perform the scan for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* For GCA group:

  1. Adults ≥ 50 years at the time of enrolment
  2. Meets 2022 American College of Rheumatology/EULAR classification criteria for giant cell arteritis
  3. Imaging evidence of active LV-GCA in the previous 4 weeks
  4. Will be managed with corticosteroid monotherapy by the standard care team.

For BCMID group:

1. Adults ≥ 18 years at the time of enrolment
2. Meets criteria for a diagnosis of a B-cell mediated immune disorder
3. Considered to have active disease by referring team
4. Will be managed as per standard of care by referring team

For AA group:

1. Adults ≥ 50 years at the time of enrolment
2. Imaging evidence of atherosclerotic aortic aneurysm

Exclusion Criteria:

1. Participants receiving corticosteroids for >4 weeks immediately prior to baseline
2. Previous diagnosis of GCA
3. History of any major morbidity which the clinical investigator considers contraindicated to study entry
4. Pregnancy or breastfeeding
5. Advanced renal dysfunction (eGFR <15ml/min/1.73m2)
6. Patients without mental capacity or willingness to provide informed consent
7. Inability or unwillingness to comply with the radiation protection advice

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For GCA group:
  1. Adults ≥ 50 years at the time of enrolment
  2. Meets 2022 American College of Rheumatology/EULAR classification criteria for giant cell arteritis
  3. Imaging evidence of active LV-GCA in the previous 4 weeks
  4. Will be managed with corticosteroid monotherapy by the standard care team.
  For BCMID group:
  1. Adults ≥ 18 years at the time of enrolment
  2. Meets criteria for a diagnosis of a B-cell mediated immune disorder
  3. Considered to have active disease by referring team
  4. Will be managed as per standard of care by referring team
  For AA group:
  1. Adults ≥ 50 years at the time of enrolment
  2. Imaging evidence of atherosclerotic aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Quantification of vascular 89Zr-RTX uptake | 0-4 months
  Quantification of vascular 89Zr-RTX uptake compared between:
  A) those with LV-GCA before and after treatment with steroids B) those with LV-GCA and a control group

SECONDARY OUTCOMES:
Correlation between vascular 89Zr-RTX uptake and peripheral blood B cell populations | 0-4 months
Correlation between vascular 89Zr-RTX uptake and temporal artery B cell populations | 0-4 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, City of Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No